CLINICAL TRIAL: NCT01487174
Title: A Multi-Center, Phase 3, Double-Blind, Randomized, and Controlled Trial of KD019 vs Erlotinib in Subjects With Stage IIIB/IV Non-Small Cell Lung Cancer Who Have Progressed After First- or Second-Line Chemotherapy
Brief Title: KD019 Versus Erlotinib in Subjects With Stage IIIB/IV Non Small Cell Lung Cancer With Progression After First- or Second-Line Chemotherapy
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Kadmon has made a business decision to terminate the study due to slow enrollment. Note the decision to terminate the study was not related to safety issues
Sponsor: Kadmon Corporation, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KD019-301
Record Dates: First submitted 2011-12-02; First posted 2011-12-07 (Estimated); Last update posted 2022-05-13 (Actual); Status verified 2022-05

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — XL647; Erlotinib Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- KD019 (Experimental): KD019 will be administered orally once daily at a dose of 300 mg. One dose reduction to 200 mg will be permitted.
  Interventions: Drug: KD019
- Erlotinib (Active Comparator): Erlotinib will be administered orally once daily at a dose of 150 mg. One dose reduction to 100 mg daily will be permitted.
  Interventions: Drug: Erlotinib

INTERVENTIONS:
Drug: KD019 — KD019 will be administered orally once daily at a dose of 300 mg. One dose reduction to 200 mg will be permitted.
  Other Names: XL647
  Arms: KD019
Drug: Erlotinib — Erlotinib will be administered orally once daily at a dose of 150 mg. One dose reduction to 100 mg daily will be permitted.
  Other Names: Tarceva
  Arms: Erlotinib

SUMMARY:
This study involves treatment with KD019 or erlotinib in patients with Non-small cell lung cancer (NSCLC) who have progressed after first- or second- line chemotherapy. It is hypothesized that KD019 can prolong survival compared with erlotinib.

ELIGIBILITY:
For Eligibility subjects must have:

* failed one or two previous courses of therapy.
* have no active brain metastasis. Treated non-active brain metastasis are acceptable.
* cannot have received an Epidermal Growth Factor Receptors inhibitor (Tarceva [erlotinib] or Iressa [gefitinib]) in the past.
* has demonstrated progressive disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2011-12-14; Primary Completion 2013-07-25 (Actual); Study Completion 2013-07-25 (Actual)

PRIMARY OUTCOMES:
Overall survival | Will be performed until documentation of progressive disease per RECIST or death due to any cause, an expected average of approximately 1year

SECONDARY OUTCOMES:
Progression-free survival | Will be performed until documentation of progressive disease per RECIST or death due to any cause, an expected average of approximately 1year
Number and type of adverse events related to KD019 | Will be performed until documentation of progressive disease per RECIST or death due to any cause, an expected average of approximately 1year
  For the purpose of data collection, all untoward events that occur after informed consent through 30 days after last dose of study treatment are to be recorded.
Objective response rate | Will be performed until documentation of progressive disease per RECIST or death due to any cause, an expected average of approximately 1year

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Yale Cancer Center, New Haven, Connecticut
  - San Juan Oncology Associates, Farmington, New Mexico